CLINICAL TRIAL: NCT00515372
Title: Depression Treatment and Screening in Ovarian Cancer Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Lance Armstrong Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID02-258; NCI-2012-02127 (Registry Identifier: NCI CTRP); 1CF2002-0000832 HM 01 (Other Grant/Funding Number: Lance Armstrong Foundation); K07CA093512-01A2 (NIH)
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Depression; Telephone Counseling; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Weekly phone calls lasting about 30 minutes. Lists of professional resources and referral recommendations will be provided.
  Interventions: Other: Telephone Counseling
- Usual Care Group (Other): Lists of professional resources and referral recommendations will be provided.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Telephone Counseling — Weekly phone calls lasting about 30 minutes.
  Other Names: Survey
  Arms: Intervention Group
Other: Usual Care — Lists of professional resources and referral recommendations will be provided.
  Arms: Usual Care Group

SUMMARY:
The goal of this behavioral research study is to find a quick and effective way to identify depression in patients with ovarian, peritoneal, or fallopian tube cancer. Another goal of this study is to compare an intervention program with "enhanced" standard care to see which may be more effective in improving quality of life for these patients.

DETAILED DESCRIPTION:
Study Participation:

If you agree to take part in this study, you will fill out a questionnaire, complete an interview (called a SCID interview), and information will be collected from your medical record.

For the questionnaire, you will answer questions about your mood, ability to cope with cancer, thoughts about cancer, and demographic information (such as your age and race). It should take between 30 and 40 minutes to complete the questionnaire.

For the SCID interview (which may be conducted during your routine visit at M. D. Anderson or by telephone), a trained interviewer will ask you questions related to the degree of depression you may be experiencing. It should take between 30 and 40 minutes to complete the SCID interview. The study staff will also show you TAT cards, which are standardized psychological testing cards, and ask you to give responses to the cards.

Information collected from your medical record will include the cancer stage, if the disease has gotten worse, treatment, and side effects. This information will help researchers learn how specific treatments affect patients.

* You may also be asked to have an informal interview on your personal experience about matters not related to depression. Information learned from this interview may need to be addressed in order to help you cope with your personal cancer experiences (such as communicating with your study doctor and study staff, financial counseling, and spiritual guidance).
* If you are not found to be eligible for the intervention group, you will be contacted again in 4 months to complete a second questionnaire and SCID interview. Both will be the same as the first questionnaire and SCID interview, except that the questionnaire will have additional questions about the type of psychosocial help you may have received outside of this research study during the 4-month period.

Study Group Randomization:

If your answers to the first questionnaire show that you might benefit from psychosocial support, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups (an intervention group or an enhanced standard care group).

Intervention Group:

If you are assigned to the intervention group, you will receive intervention plus enhanced standard care that is described below. For the intervention, you will have 10 telephone calls by a trained psychologist under the supervision of a licensed psychiatrist. The psychologist will discuss with you and teach you cognitive-behavioral techniques. These techniques will show you ways to relax, how to schedule physical activities, and how to identify and counter negative thoughts. You will also receive a journal to write down ideas on how to practice fighting depression. These intervention calls will last about 30 minutes each time, and will occur once a week (almost every week).

Standard Care Group:

If you are assigned to the enhanced standard care group, you will be informed of the results of the analysis of your first questionnaire and provided with a list of professional resources and referral recommendations for psychosocial counseling. Your treating doctor and/or regular doctor will also be informed of these results as well. After 4 months in this group, you will be able to receive the intervention as described above.

Additional Information:

In order to check for quality control (to see if the intervention and SCID interview have been appropriately done), a random sample of telephone counseling sessions (from the intervention group) will be tape recorded, and a random sample of interviews (the SCID interviews) will be tape recorded and/or videotaped. Before any information is tape recorded and/or videotaped, you will be asked for your permission.

The tape recording and/or videotaping will be done by members of study staff. No identifying information (such as your name and medical record number) will be recorded on the audiotape and/or videotape. The audiotape and/or videotape will only be labeled with study ID numbers.

Length of Study:

If your answers to the first questionnaire do not show that you might benefit from psychosocial support, your participation will be over (in about 4 months) after you have completed the follow-up questionnaire and SCID interview.

If you are assigned to the intervention, your participation will be over (in about 4 months) once you have completed the 10 weekly intervention sessions.

If you are assigned to the standard care group, your participation will be over in about 4 months, or about 8 months if you are able to also take part in the intervention once you have completed your participation in the standard care group.

This is an investigational study. Up to 588 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women are eligible if they a) are on active treatment, but not at the end of a treatment regimen) for newly diagnosed, recurrent, or persistent ovarian cancer or peritoneal cancer or fallopian tube cancer (any stage) c) are at least 18 years of age; d) speak and read English at a 7th grade level; e) are oriented to time, person, and place; g) have a Zubrod performance status (49) of 0-2; and h) provide informed consent.
2. They are eligible for the pilot intervention phase of the study if they have a diagnosis of major depressive disorder, dysthymic disorder, adjustment disorder with depressed mood, minor depression, major depression in partial remission, or recurrent brief depressive disorder.

Exclusion Criteria:

1) They will be excluded from this phase of the study if they are diagnosed as having a bipolar disorder or psychosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2002-12-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Responses to Questionnaire Assessment of Depression Measures | Baseline assessment repeated at four months, and completion of first chemotherapy regimen for newly diagnosed ovarian, peritoneal, or fallopian tube cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H. Shinn, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org